CLINICAL TRIAL: NCT05895123
Title: Comparative Study Between the Effects of High Doses Rosuvastatin and Atorvastatin on Ventricular Remodeling in Patients With ST-Segment Elevation Myocardial Infarction
Brief Title: Comparison Between the Effects of High Doses Statin on Ventricular Remodeling in STEMI Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Damanhour University (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: statinstudy
Record Dates: First submitted 2022-10-11; First posted 2023-06-08 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: ST-segment Elevation Myocardial Infarction
Keywords: Statin; remodeling; STEMI
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Rosuvastatin Calcium; Atorvastatin; ORANGE protein, Arabidopsis

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rosuvastatin group (Experimental): patients will receive Rosuvastatin orally (20 mg) at night once daily
  Interventions: Drug: Rosuvastatin 20 mg
- Atorvastatin group (Experimental): patients will receive Atorvastatin orally (40 mg) at night once daily
  Interventions: Drug: Atorvastatin 40mg

INTERVENTIONS:
Drug: Rosuvastatin 20 mg — patients will receive one tablet rosuvastatin 20 mg every night
  Other Names: cholerose
  Arms: Rosuvastatin group
Drug: Atorvastatin 40mg — patients will receive one tablet Atorvastatin 40 mg every night
  Other Names: ator
  Arms: Atorvastatin group

SUMMARY:
STEMI is a serious type of coronary heart disease, which is a major cause of disability and death. Morphologically the key feature of remodeling is myocyte hypertrophy, myocyte loss from necrosis or apoptosis, as well as interstitial cell growth especially fibroblast proliferation leading to myocardial fibrosis .

Elevated serum LDL-cholesterol concentrations play a proatherogenic role by stimulating inflammation and oxidative processes.

Statins have been documented to retard fibrosis and ventricular hypertrophy by the cessation of myofibroblast activity. Clinical studies have proven that statins not only regulate lipids but also improve myocardial fibrosis, regulate cell proliferation and apoptosis, regulate ventricular remodeling, and protect the myocardium

DETAILED DESCRIPTION:
1. Ethical committee approval will be obtained from Ethics committee of Faculty of Pharmacy, Damanhour University.
2. All participants should agree to take part in this clinical study and will provide informed consent.
3. (80) patients diagnosed with STEMI will be enrolled from Alexandria university hospital.
4. Serum samples will be collected from patients at the time of admission for measuring the biomarkers.
5. Echocardiogram also will be obtained at the time of admission.
6. All enrolled patients will be divided into two group to receive either Atorvastatin (40 mg) or Rosuvastatin (20mg).
7. All patients will be followed up during 3 months' period. At the end of 3 months, Serum samples will be collected from patients for measuring the biomarkers and Echocardiogram will be repeated.
8. Statistical tests appropriate to the study design will be conducted to evaluate the significance of the results.
9. Results, conclusion, discussion, and recommendations will be given.

ELIGIBILITY:
Inclusion Criteria:

1. Electrocardiogram showed abnormal elevation of the ST segment.
2. First myocardial infarction occurred.
3. The patients received one-stage percutaneous coronary intervention (PCI) therapy within 12 h.

Exclusion Criteria:

1. Severe cardiac insufficiency.
2. Hepatic insufficiency (continuous increase of serum transaminase more than 3 times of the upper limit of normal level).
3. Renal insufficiency (creatinine clearance rate <30 mL/min).
4. Addition of others blood lipid lowering and antioxidant drugs during follow up period.
5. Familial hypercholesterolemia.
6. Malignant tumor.
7. Immune system disease.
8. Acute infectious disease.
9. Hypersensitivity to rosuvastatin and Atorvastatin.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of the effect on ventricular remodeling | 3 months
  MMP9,sST2 and CRP level will be measured and monitoring the change in their levels Echocardiogram will be obtained and monitoring the change in echocardiogram indexes.

SECONDARY OUTCOMES:
Evaluation of the effect on lipid parameters and liver enzymes | 3 months
  lipid parameters and liver enzymes level will be measured and monitoring the change in their levels

CONTACTS AND LOCATIONS:
Overall Officials: Zeinab M Elhadad, bachelor, Principal Investigator — demonstrator of Clinical Pharmacy, Damanhour University.; Amira B Kassem, PhD, Study Director — Lecturer of Clinical Pharmacy, Damanhour University.; Ahmed salahaldin, PHD, Study Director — Lecturer of biochemisrty, Damanhour University.; noha ahmad, PHD, Study Chair — Lecturer of Clinical Pharmacy, Damanhour University.; ahmad alamrawy, PHD, Study Chair — Lecturer of cardiology , Faculty of medicine, Alexandria University.
Locations (1):
- Damanhour University, Damanhūr, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khurana S, Gupta S, Bhalla H, Nandwani S, Gupta V. Comparison of anti-inflammatory effect of atorvastatin with rosuvastatin in patients of acute coronary syndrome. J Pharmacol Pharmacother. 2015 Jul-Sep;6(3):130-5. doi: 10.4103/0976-500X.162011. PMID 26311995
- [Background] Sutton MG, Sharpe N. Left ventricular remodeling after myocardial infarction: pathophysiology and therapy. Circulation. 2000 Jun 27;101(25):2981-8. doi: 10.1161/01.cir.101.25.2981. No abstract available. PMID 10869273
- [Background] Reddy R, Chahoud G, Mehta JL. Modulation of cardiovascular remodeling with statins: fact or fiction? Curr Vasc Pharmacol. 2005 Jan;3(1):69-79. doi: 10.2174/1570161052773915. PMID 15638784
- [Background] Berezin AE, Berezin AA. Adverse Cardiac Remodelling after Acute Myocardial Infarction: Old and New Biomarkers. Dis Markers. 2020 Jun 12;2020:1215802. doi: 10.1155/2020/1215802. eCollection 2020. PMID 32626540
- [Background] Neri M, Riezzo I, Pascale N, Pomara C, Turillazzi E. Ischemia/Reperfusion Injury following Acute Myocardial Infarction: A Critical Issue for Clinicians and Forensic Pathologists. Mediators Inflamm. 2017;2017:7018393. doi: 10.1155/2017/7018393. Epub 2017 Feb 13. PMID 28286377
- [Derived] Elhadad ZM, Kassem AB, Amrawy AME, Salahuddin A, El-Bassiouny NA. Comparative Study Between the Effects of High Doses of Rosuvastatin and Atorvastatin on Ventricular Remodeling in Patients with ST-Segment Elevation Myocardial Infarction. Cardiovasc Drugs Ther. 2025 Oct;39(5):1113-1123. doi: 10.1007/s10557-024-07621-w. Epub 2024 Sep 12. PMID 39264503
- See also: Luo R, Sun X, Shen F, Design BH-D, Development undefined, 2020 undefined. Effects of High-Dose Rosuvastatin on Ventricular Remodelling and Cardiac Function in ST-Segment Elevation Myocardial Infarction. ncbi.nlm.nih.gov [Internet]. [cited 2021 Aug 20]; — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7520152/